CLINICAL TRIAL: NCT02721485
Title: Crystalloid FLUID Choices for Resuscitation of Hospital Patients: A Pragmatic Cluster Cross Over Pilot Trial
Brief Title: Crystalloid FLUID Choices for Resuscitation of Hospital Patients
Acronym: FLUID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20150619-01H
Record Dates: First submitted 2016-01-18; First posted 2016-03-29 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Fluid Therapy
Keywords: Ringer's Lactate; Normal Saline; resuscitation fluids; hypovolemia
MeSH Terms: conditions — Hypovolemia | interventions — Ringer's Lactate; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline (Other): Half of the hospitals will be allocated to start the 90-day test period using Normal Saline administered as 500 or 1000 ml boluses or infusions as specified by the treating physicians. After a 1 week run out, half of participating hospitals will have up to 2 weeks to switch out stock then will be crossed over to using Ringer's Lactate following a 1 week run in as 500 or 1000 ml boluses or infusions as specified by the treating physicians for the final 90-day test period.
  Interventions: Other: Ringer's Lactate
- Ringer's Lactate (Other): Half of the hospitals will be allocated to start the 90-day test period using Ringer's Lactate administered as 500 or 1000 ml boluses or infusions as specified by the treating physicians. After a 1 week run out, half of participating hospitals will have up to 2 weeks to switch out stock then will be crossed over to using Normal Saline following a 1 week run in as 500 or 1000 ml boluses or infusions as specified by the treating physicians in for the final 90-day test period.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Other: Ringer's Lactate — After a 1 week run in half of participating hospitals will be crossed over to using Ringer's Lactate as 500 or 1000 ml boluses or infusions as specified by the treating physicians for the second 90-day test period.
  Arms: Normal Saline
Other: Normal Saline — After a 1 week run in half of participating hospitals will be crossed over to using Normal Saline as 500 or 1000 ml boluses or infusions as specified by the treating physicians for the final 90-day test period.
  Arms: Ringer's Lactate

SUMMARY:
Salt fluids are used extensively for acutely ill patients who are admitted to hospital. Two salt fluids commonly used are Normal Saline and Ringer's Lactate. Both are used to rehydrate patients, restore fluid volume and help stabilize blood pressure and failing organs. Both salt fluids have been used for several decades. Until recently, it was thought the fluids are essentially equivalent other than some minor differences related to the concentration of salt components (sodium and chloride) and buffers (Ringer's Lactate has lactate as a buffer). Recent data suggest that salt fluids containing less chloride like the Ringer's Lactate, cause less acid in the blood, less kidney failure, and less death. However, the studies to date are small and weak in their design and it is possible that there are no important differences that affect patients. Hence, the research team will conduct a robust pragmatic clinical trial where several academic and community hospitals will be randomized to use either Ringer's Lactate only or Normal Saline only for a period of three months. The trial will yield high quality and robust data to determine if Ringers Lactate reduces death and re-admissions to hospital. Before embarking on this large-scale trial, it is important to conduct a smaller (pilot) trial to evaluate if the larger trial will be feasible and not too costly. In this small trial involving no less than 4 hospitals, the investigators will determine how well the fluid interventions are adhered to in each hospital, record how long it takes to receive approval from research ethics boards and be ready to start the study. The investigators will also record challenges and develop solutions related to the operations of the trial, and describe important clinical and outcome data essential for the design and planning of the large trial.

DETAILED DESCRIPTION:
Other than the administration of oxygen, crystalloid resuscitation fluids are the most common intervention administered to the majority of hospitalized patients. These fluids may be used as a life saving measure to re-establish hemodynamic stability, for rehydration, and to replace losses and maintain intravascular volume in the surgical setting. In the province of Ontario alone, approximately 1 million patients per year will receive one or both of these resuscitation fluids during their hospital admission. The two most common usual care resuscitation crystalloid fluids are Normal Saline and Ringer's Lactate and until recently there was no evidence to suggest that one crystalloid fluid was clinically superior to the other. However, the safety of Normal Saline is now being questioned due to its high chloride content and its association with the development of hyperchloremic metabolic acidosis. Studies in healthy volunteers and observational studies in the critically ill and surgical patient populations have associated saline with an increased risk of acute renal injury and requirement for dialysis, post-operative infections, death and increased resource and blood transfusion use. The evidence base is currently weak given that the majority of studies are observational and suffer from methodological weaknesses including confounding by indication, selection bias, and inability to disentangle the effects of a specific fluid due to interaction of co-interventions administered. As such, several authors and editorials have called for adequately powered randomized controlled trials with clinically relevant outcomes to determine if Ringer's Lactate is indeed superior to Normal Saline for resuscitation.

Given their widespread use, small differences in clinical outcomes between crystalloid resuscitation fluids are highly relevant. Furthermore, small absolute differences in important clinical outcomes translate into significant savings to hospitals and the health care system. To illustrate, if death and hospital re-admissions were each reduced by an absolute 0.5%, this would translate to approximately 2500 lives saved and savings of 10 million dollars to the Ontario health care system. Hence, in collaboration with the Canadian Critical Care Trials Group, the Crystalloid FLUID Choices for Hospitalized Patients (FLUID) trial will examine whether Ringer's Lactate as compared to Normal Saline reduces clinically important outcomes such as death, and hospital re-admissions - outcomes that are particularly relevant to hospitals and the health care system. This proposal is a large pragmatic cluster cross-over comparative effectiveness trial that will be conducted in both academic and community centres in Ontario. It will involve waivers of consent and a novel design making use of provincially available health administrative data through the Institute of Clinical Evaluative Sciences (ICES) to facilitate all data collected in the trial. The trial will answer this fundamental fluid resuscitation question with much less cost in comparison to an individual patient randomized controlled trial. It will help build expertise and capacity for future trials of similar design in the province of Ontario and throughout Canada. However, prior to embarking on a large-scale trial, it is imperative to conduct a pilot trial to determine feasibility and optimize the trial design.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the participating hospitals for the first time in the last 90 days (index admission) over the duration of the study period.

Exclusion Criteria:

* Neonates (< 30 days)
* Physicians may also opt out of the use of the allocated study fluid for individual patients if there is a strong preference to do so.

Ages: 30 Days to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30000 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-01-13 (Actual); Study Completion 2018-01-13 (Actual)

PRIMARY OUTCOMES:
Feasibility: adherence to protocol | Up to six months
  Compliance defined as at least 80% of the prescribed study fluid being administered in the participating hospitals over the 2, 3-month study periods.
Feasibility: time to research ethics board approval | Up to three months
  Compliance defined as taking no longer than 3 months to achieve
Feasibility: readiness to initiate protocol | Up to three months
  Compliance defined as taking no longer than 3 months after ethics approval

CONTACTS AND LOCATIONS:
Overall Officials: Lauralyn McIntyre, MD MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (4):
- Canada (4):
  - Hamilton General Hospital, Hamilton, Ontario
  - Ottawa Hospital Civic Campus, Ottawa, Ontario
  - The Ottawa Hospital General Campus, Ottawa, Ontario
  - Queensway Carleton Hosptial, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No
This is a cluster-randomized crossover study, with the hospital as the unit of randomization. Individual patient data will not be collected.

REFERENCES:
- [Derived] McIntyre LA, Fergusson DA, McArdle T, Fox-Robichaud A, English SW, Martin C, Marshall J, Cook DJ, Graham ID, Hawken S, McCartney C, Menon K, Saginur R, Seely A, Stiell I, Thavorn K, Weijer C, Iyengar A, Muscedere J, Forster AJ, Taljaard M; Canadian Critical Care Trials Group. FLUID trial: a hospital-wide open-label cluster cross-over pragmatic comparative effectiveness randomised pilot trial comparing normal saline to Ringer's lactate. BMJ Open. 2023 Feb 3;13(2):e067142. doi: 10.1136/bmjopen-2022-067142. PMID 36737087
- [Derived] McIntyre L, Taljaard M, McArdle T, Fox-Robichaud A, English SW, Martin C, Marshall J, Menon K, Muscedere J, Cook DJ, Weijer C, Saginur R, Maybee A, Iyengar A, Forster A, Graham ID, Hawken S, McCartney C, Seely AJ, Stiell IG, Thavorn K, Fergusson DA. FLUID trial: a protocol for a hospital-wide open-label cluster crossover pragmatic comparative effectiveness randomised pilot trial. BMJ Open. 2018 Aug 23;8(8):e022780. doi: 10.1136/bmjopen-2018-022780. PMID 30139908